CLINICAL TRIAL: NCT05816005
Title: Performance of Whole Body MRI in Extraplevic Disease Detection in Patients Undergoing Pelvic Exenteration for Gynecological Maligniancies
Acronym: WHOLE BODY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3813
Record Dates: First submitted 2023-03-29; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective observational diagnostic study is to investigate the diagnostic accuracy od extrapelvic disease detection using Whole-body-MRI (WB-MRI) in patients with gynecologic cancer candidate to the pelvic exenteration.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Written Informed Consent
* All patients with recurrent gynecological cancer that are planned to undergo pelvic exenteration or laterally extended pelvic resection, both with curative and palliative intent
* Patients considered fit for srugery

Exclusion Criteria:

* Controindication to MRI (Claustrophobia, implanted ferromagnetic materials or foreign objects, Known intolerance or controindication to the MRI contrast agent, cardiac pacemaker)
* Individuals who are not able or willing to tolerate the required prologed stationary supine position during examination (approximately 40-60 minutes)
* Patient unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women can be included
Study Population: Patients with pelvic maligniancies that will undergo to preoperative contrast enhanced MRI to precisely define the extent of local and/or distant disease before pelvic exenteration
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of diagnostic accuracy for extrapelvic disease detection using whole-body MRI | Through study completion, an average of 2 yearS

SECONDARY OUTCOMES:
Agreement between WB-MRI and PET-CT in detecting extrapelvic involvement | Through study completion, an average of 2 yearS

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitaro "A. Gemelli" IRCCS, Roma, Italy